CLINICAL TRIAL: NCT06026059
Title: Interest of a Visual Scale for Evaluating Food Portions as a Screening Tool for Nutritional Risk in Pediatrics
Acronym: EFImôme
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0059
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Undernutrition
Keywords: undernutrition; diagnostic; screening
MeSH Terms: conditions — Malnutrition; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- interview with the dietician: Initially, parent(s) and child will be interviewed together, details of the dietary record, as well as the data needed to calculate the nutritional risk score will be obtained.
  The interview will then be only with the child, he will be asked to determine, on his/her own, the portion of food he/she thinks he/she ate the previous evening, using the SEFI score.
  Finally, one of the two parents will determine, on their own, the portion of food they think their child ate the previous evening, using the SEFI score.

SUMMARY:
In current practice, there are various nutritional risk scores and diagnostic tools which are used in both inpatient and outpatient settings,however, in some cases, these tools cannot be used due to lack of data.

That's why a tool that doesn't require any anthropometric parameters, such as a visual food intake scale, could be useful to for medical and paramedical staff. In this way, a larger proportion of the paediatric population could benefit from nutritional screening.

DETAILED DESCRIPTION:
HAS defines undernutrition as a state of nutritional imbalance, characterized by a negative energy and/or protein balance. This negative balance may be linked to a deficit in isolated intake and/or an increase in energy and/or protein expenditure.

In current practice, there are various nutritional risk scores and diagnostic tools which are used in both inpatient and outpatient settings. Practitioners can use discs to quickly and easily determine BMI, which corresponds to the ratio of Weight (Kg) / Height² (m). However, in some cases, these tools cannot be used due to lack of data.

That's why a tool that doesn't require any anthropometric parameters could be useful to for medical and paramedical staff. In this way, a larger proportion of the paediatric population could benefit from nutritional screening.

In adults, a visual food intake scale exists and has been validated for screening for nutritional risk. The hypothesis of this study is that the visual food intake scale could be a good tool for screening for nutritional risk in paediatrics

ELIGIBILITY:
Inclusion Criteria:

* Child able to be weighed and measured
* Family with Internet access and telephone number
* Child and at least one parent present during day hospitalization,
* Child able to respond to the SEFI® scale and having completed the 3-day food intake at home

Exclusion Criteria:

* Children and/or parents with comprehension and/or communication difficulties
* Children with any pathological condition making interpretation of results difficult from the investigator's point of view
* Children receiving nutritional support: enteral and parenteral nutrition.
* Child with nutritional follow-up

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a scheduled hospitalization, according to the day hospital scheduling list, will be proposed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the SEFI scale as a screening tool for child's nutritional risk. | Day 1
  The correlation between the self evaluation of food intake (SEFI) scale, with scores from 0 to 10, indicating the presence of malnutrition score if score is inferior to 7 or absence of malnutrition if score superior to 7/10, and the STRONGkids score will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Céline BARDE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No